CLINICAL TRIAL: NCT06366191
Title: Psychotrauma Prevention Algorithm : Randomized, Controlled Pilot Study
Acronym: A2P
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/CHU/08
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Psychological Trauma
MeSH Terms: conditions — Psychological Trauma | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prevention algorithm (Experimental): Patient will have the current support for psychotrauma and psychotrauma prevention algorithm.
  Interventions: Other: prevention algorithm
- Current support for psychotrauma (Active Comparator): Patient will have the current support for psychotrauma.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: prevention algorithm — a health watch adapted to stress and dissociative symptoms
  Arms: Prevention algorithm
Other: Standard care — Standard care for post traumatic stress disorder
  Arms: Current support for psychotrauma

SUMMARY:
A randomized pilot study which proposes to patients having suffered a traumatic event to have either only the standard care or the standard care associated with adaptated psychotrauma watch and prevention system.

ELIGIBILITY:
Inclusion Criteria:

* Person who the vital prognosis has or could have been committed or having felt a threat to his physical and/or psychological integrity
* After a potentially traumatic event dating from a minimum of 72 hours to a maximum of 1 week
* for which the CUMP or the psychotrauma regulation platform has been requested
* having lived or being a direct witness of the event
* knowing how to read and write
* affiliate or beneficiary of a social security scheme
* having signed a consent

Non-inclusion Criteria:

* guardianship or curatorship
* unable to receive phone calls
* unable to go to a place for consultation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
study acceptability rate | 6 months after inclusion
  Number of included patient divided by number of patients to whom the study was offered.
  Study acceptability rate of 50% is expected.

SECONDARY OUTCOMES:
Adherence of patient to the watch | 1 month after inclusion
  Number of patient contacted by phone having completed the scales divided by number of patient contacted.
Adherence of patient to the health watch | 3 months after inclusion
  Number of patient contacted by phone having completed the scales divided by number of patient contacted
Patient satisfaction (quantitatif) | 3 months after inclusion
  A questionnaire will be completed by the patient
Patient satisfaction (qualitatif) | 3 months after inclusion
  semi-structured interview carried-out in 3 patients volunteers (45 minutes)
Strong points of the health watch | 3 months after inclusion
  semi-structured interview carried-out in volunteer caregivers (doctor, nurse, psychologist)
Evolution of the patient journey in experimental arm | 3 months after inclusion
  number an percentage of patient who have changed watch
Occurrence of post-traumatic stress disorder | 3 months after inclusion
  Evaluation by Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5). Score between 0 and 80. Score < 38 : no post-traumatic stress disorder Score = or > 38 : post-traumatic stress disorder
Complications associated with post-traumatic stress disorder | at inclusion
  assessed by C-SSRS (Columbia-Suicide Severity Rating Scale). Assessment of suicide risk in patient. No score for this scale.
Complications associated with post-traumatic stress disorder | 3 months after inclusion
  assessed by C-SSRS (Columbia-Suicide Severity Rating Scale). Assessment of suicide risk in patient. No score for this scale.
Complications associated with post-traumatic stress disorder | 3 months after inclusion
  assessed by the Hospital Anxiety and Depression Scale (HADS). 1 subscore for anxiety scale (HADS-A) between 0 and 21
  1 subscore for depression scale (HADS-D) between 0 and 21 Overall score between 0 and 42 HADS-A + HADS-D scores). Score < or = 7 : no symptom Score = or > 8 : symptom the higher the score, the more severe the symptoms
Complications associated with post-traumatic stress disorder | 3 months after inclusion
  assessed by WHO Quality of life - Bref (WHOQOL Bref). This scale assessed 4 domains : physical health, mental health, social relations and the environment.
  Overall Score is between 26 and 130. the higher the score, the better the quality of life